CLINICAL TRIAL: NCT00316030
Title: A Phase I Study of Bexarotene in Patients With Acute Myeloid Leukemia
Brief Title: Study of Bexarotene in Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Donald Tsai, M.D., University of Pennsylvania
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 12403; 708935
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2008-03

CONDITIONS: AML; Acute Myeloid Leukemia
Keywords: AML; Acute Myeloid Leukemia; Bexarotene; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Bexarotene

INTERVENTIONS:
Drug: Bexarotene

SUMMARY:
Bexarotene may be useful in the treatment of Acute Myeloid Leukemia (AML). This is the first study on the use of bexarotene to treat patients with AML. The main purpose of this study is to establish the proper dose of bexarotene when used to treat AML. The side effect profile of bexarotene in patients with AML will also be explored.

DETAILED DESCRIPTION:
Despite recent advances in cancer treatment, the prognosis is still poor for patients with relapsed or chemotherapy resistant AML. Further aggressive chemotherapy can be attempted, but generally yields poor results. This clinical study is the first use of bexarotene in the treatment of patient with relapsed or chemotherapy resistant AML. The main purpose of the study is to identify the maximum safe dose of bexarotene in patient with AML. Another objective of the study is to explore the side effect profile of bexarotene in AML patients. The study is organized so that the initial patients will get a low dose of bexarotene to be taken daily. If these patients tolerate the drug, then later patients will get higher daily doses. Further groups of patients will continue to increase their dose of bexarotene until a maximum tolerated dose is identified. The stu dy will end at that point. Patients will take the drug daily by mouth until such a time that their AML is worsening or they are experiencing unacceptable side effects. Their participating will end at that point.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Must have a histologically confirmed diagnosis of non-M3 AML as proven by bone marrow biopsy. Patients with CML in myeloid blast crisis are eligible.
* Willing and able to give informed consent.
* Must have received prior induction therapy with conventional chemotherapy and/or Mylotarg or otherwise not be eligible for conventional chemotherapy
* ECOG performance status of 0-2
* Must have recovered from the toxicities of prior chemotherapy.
* Women of childbearing potential must use effective contraception after enrollment in this study and have a negative pregnancy test within 1 week of study enrollment. They must continue to use effective contraception for 3 months after stopping bexarotene.
* Men must agree to use effective methods of contraception while taking bexarotene and for 3 months after stopping therapy.

Exclusion Criteria:

* History of pancreatitis.
* Active alcohol abuse
* Taken bexarotene in the past.
* WBC >10,000/uL at the time of enrollment. Patients may be taking hydrea for WBC control at the time of enrollment.
* Cytotoxic chemotherapy or Mylotarg within the past 7 days other than hydrea.
* Significant organ dysfunction: total bilirubin>3x ULN, AST or ALT>3x ULN, creatinine>4mg/dL, on blood pressure supporting medications or mechanical ventilation.
* Serious medical or psychiatric conditions that may compromise the safety of the patient while participating in this study.
* Women of childbearing potential who are pregnant or actively breast feeding.
* Active participant in any other investigational treatment study for their AML.
* Unable/unwilling to perform required follow-up.
* Life expectancy of less than 1 month.
* Use of blood growth factors (G-CSF, GM-CSF, Aranesp, erythropoietin, or Neumega) within 1 week prior to treatment initiation.
* Uncontrolled hyperlipidemia (triglycerides>1000 while on treatment with triglyceride lowering medications).
* History of myeloablative allogeneic stem cell transplant.
* Known history of HIV.
* Uncontrolled active infection
* Known active CNS involvement with AML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Start 2004-01

PRIMARY OUTCOMES:
To identify the maximum tolerated daily dose of bexarotene in patients with Acute Myeloid Leukemia
To assess the toxicities of bexarotene in patients with AML

CONTACTS AND LOCATIONS:
Overall Officials: Donald E Tsai, M.D., Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Boehm MF, Zhang L, Badea BA, White SK, Mais DE, Berger E, Suto CM, Goldman ME, Heyman RA. Synthesis and structure-activity relationships of novel retinoid X receptor-selective retinoids. J Med Chem. 1994 Sep 2;37(18):2930-41. doi: 10.1021/jm00044a014. PMID 8071941
- [Background] Boehm MF, Zhang L, Zhi L, McClurg MR, Berger E, Wagoner M, Mais DE, Suto CM, Davies JA, Heyman RA, et al. Design and synthesis of potent retinoid X receptor selective ligands that induce apoptosis in leukemia cells. J Med Chem. 1995 Aug 4;38(16):3146-55. doi: 10.1021/jm00016a018. PMID 7636877
- [Background] Kizaki M, Dawson MI, Heyman R, Elster E, Morosetti R, Pakkala S, Chen DL, Ueno H, Chao W, Morikawa M, Ikeda Y, Heber D, Pfahl M, Koeffler HP. Effects of novel retinoid X receptor-selective ligands on myeloid leukemia differentiation and proliferation in vitro. Blood. 1996 Mar 1;87(5):1977-84. PMID 8634447
- [Background] Asou H, Koike M, Elstner E, Cambell M, Le J, Uskokovic MR, Kamada N, Koeffler HP. 19-nor vitamin-D analogs: a new class of potent inhibitors of proliferation and inducers of differentiation of human myeloid leukemia cell lines. Blood. 1998 Oct 1;92(7):2441-9. PMID 9746784
- [Background] Esteva FJ, Glaspy J, Baidas S, Laufman L, Hutchins L, Dickler M, Tripathy D, Cohen R, DeMichele A, Yocum RC, Osborne CK, Hayes DF, Hortobagyi GN, Winer E, Demetri GD. Multicenter phase II study of oral bexarotene for patients with metastatic breast cancer. J Clin Oncol. 2003 Mar 15;21(6):999-1006. doi: 10.1200/JCO.2003.05.068. PMID 12637463
- [Background] Rizvi N, Hawkins MJ, Eisenberg PD, Yocum RC, Reich SD; Ligand L1069-20 Working Group. Placebo-controlled trial of bexarotene, a retinoid x receptor agonist, as maintenance therapy for patients treated with chemotherapy for advanced non-small-cell lung cancer. Clin Lung Cancer. 2001 Feb;2(3):210-5. doi: 10.3816/clc.2001.n.005. PMID 14700480
- [Background] Duvic M, Hymes K, Heald P, Breneman D, Martin AG, Myskowski P, Crowley C, Yocum RC; Bexarotene Worldwide Study Group. Bexarotene is effective and safe for treatment of refractory advanced-stage cutaneous T-cell lymphoma: multinational phase II-III trial results. J Clin Oncol. 2001 May 1;19(9):2456-71. doi: 10.1200/JCO.2001.19.9.2456. PMID 11331325
- [Background] Rizvi NA, Marshall JL, Dahut W, Ness E, Truglia JA, Loewen G, Gill GM, Ulm EH, Geiser R, Jaunakais D, Hawkins MJ. A Phase I study of LGD1069 in adults with advanced cancer. Clin Cancer Res. 1999 Jul;5(7):1658-64. PMID 10430065